CLINICAL TRIAL: NCT00784303
Title: Phase II, Multicenter, Open-label, Single Arm Trial to Evaluate the Safety and Efficacy of Oral E7080 in Medullary and Iodine-131 Refractory, Unresectable Differentiated Thyroid Cancers, Stratified by Histology
Brief Title: Evaluating the Safety and Efficacy of Oral Lenvatinib in Medullary and Iodine-131 Refractory, Unresectable Differentiated Thyroid Cancers, Stratified by Histology
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-201
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2019-03

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DTC cohort (Experimental): This arm will enroll participants with radioiodine (131 I)-refractory/resistant differentiated thyroid cancer.
  Interventions: Drug: Lenvatinib (DTC Cohort)
- MTC cohort (Experimental): This arm will enroll participants with medullary thyroid cancer.
  Interventions: Drug: Lenvatinib (MTC Cohort)

INTERVENTIONS:
Drug: Lenvatinib (DTC Cohort) — 24 mg lenvatinib (two 10 mg tablets and one 4 mg tablet) given orally, once daily, or 10 mg lenvatinib orally twice daily (20 mg total). Out of 58 participants in the DTC cohort, 56 participants received 24 mg lenvatinib once daily and 2 participants received 10 mg lenvatinib twice daily (total 20 mg daily), given continuously in 28-day treatment cycles.
  Other Names: E7080, LENVIMA
  Arms: DTC cohort
Drug: Lenvatinib (MTC Cohort) — 24 mg lenvatinib (two 10 mg tablets and one 4 mg tablet) given orally, once daily given continuously in 28-day treatment cycles.
  Other Names: E7080, LENVIMA
  Arms: MTC cohort

SUMMARY:
The purpose of this study is to determine the safety and efficacy of oral lenvatinib in participants with medullary thyroid cancer (MTC) or radioiodine (131 I)-refractory/resistant differentiated thyroid cancer (DTC), unresectable differentiated thyroid cancers, stratified by Histology.

DETAILED DESCRIPTION:
This study contained 3 Phases: the Pretreatment Phase, the Treatment Phase, and the Extension Phase. The Pretreatment Phase lasted no longer than 28 days. Informed consent was obtained and protocol eligibility and disease characteristics were established prior to treatment. The Treatment Phase consisted of a Treatment Period and a Follow-up Period. The Treatment Period of the Treatment Phase began at the time that the first participant began study drug administration and ended at the time when all participants enrolled completed 8 cycles of treatment or discontinued study treatment prior to the eighth cycle (ie, time of data cutoff for the primary study analysis [Primary Completion Date]). All participants then entered the Extension Phase. The Extension Phase consisted of a Treatment Period and a Follow-up Period. The Extension Phase began immediately after the Treatment Phase ended and included all participants that were either still receiving treatment or in follow-up. The time of data cutoff for the primary study analysis occurred when all subjects in the study completed 8 cycles of treatment or discontinued study treatment prior to the eighth cycle.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically confirmed diagnosis of medullary thyroid cancer (MTC) or differentiated thyroid cancer (DTC).
2. Measurable disease meeting the following criterion:

   1. At least one lesion (greater than or equal to 1.5 cm in longest diameter for non-lymph nodes and greater than or equal to 2.0 cm in longest diameter for lymph nodes) which is serially and accurately measurable according to modified response evaluation criteria in solid tumours (RECIST) using either computed tomography (CT) or magnetic resonance imaging (MRI).
   2. Lesions that have had electron beam radiotherapy must show evidence of progressive disease based on modified RECIST to be deemed a target lesion.
3. Evidence of disease progression by RECIST using site assessment of CT/MRI scans within 12 months (+1 month to allow for variances in patient scanning intervals) prior to study entry.
4. DTC must be 131-I refractory/resistant: never demonstrated 131-I uptake, progression despite 131-I uptake, or cumulative dose of 131-I of greater than 600 millicurie (mCi) (last dose given at least 6 months prior to study entry).
5. Well controlled blood pressure prior to study entry.

Exclusion criteria:

1. Anaplastic thyroid carcinoma, thyroid lymphoma, mesenchymal tumors of the thyroid, metastases to the thyroid.
2. Brain or leptomeningeal metastases.
3. Significant cardiovascular impairment (history of congestive heart failure, New York Heart Association [NYHA] Class II, unstable angina or myocardial infarction within 6 months of study start, or serious cardiac arrhythmia).
4. Marked baseline prolongation of QT/corrected QT (QTc) interval.
5. Proteinuria greater than 1+ or greater than 30 mg in dipstick testing.
6. Active hemoptysis (bright red blood of at least one-half teaspoon) in the 28 days prior to study entry.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-11-06 (Actual); Primary Completion 2011-04-11 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (23):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Los Gatos, California
  - Mission Viejo, California
  - Santa Monica, California
  - Torrance, California
  - Aurora, Colorado
  - Orlando, Florida
  - Tampa, Florida
  - Roswell, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - Jefferson City, Missouri
  - Lebanon, New Hampshire
  - Montclair, New Jersey
  - Houston, Texas
  - Long Beach, Washington
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (3):
  - St Leonards, New South Wales
  - Brisbane
  - Melbourne
- France (4):
  - Lyon
  - Paris
  - Reims
  - Villejuif
- Italy (6):
  - Ferrara
  - Milan
  - Naples
  - Pisa
  - Rome
  - Siena
- Poland (2):
  - Gliwice
  - Poznan
- United Kingdom (4):
  - Cardiff
  - Glasgow
  - London
  - Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 162 participants were screened for entry into the study, from which 45 were screening failures and 117 entered into the study and were treated.
Groups:
- DTC Cohort: Participants with radioiodine (131 I)-refractory/resistant differentiated thyroid cancer (DTC) received 24 mg lenvatinib (two 10 mg tablets and one 4 mg tablet) orally, once daily or 10 mg lenvatinib orally twice daily in 28-day treatment cycles. Out of 58 participants in the DTC cohort, 56 participants received 24 mg lenvatinib once daily and 2 participants received 10 mg lenvatinib twice daily (total 20 mg daily), given continuously in 28-day treatment cycles.
- MTC Cohort: Participants with medullary thyroid cancer (MTC) received 24 mg lenvatinib (two 10 mg tablets and one 4 mg tablet) given orally, once daily continuously in 28-day treatment cycles.
Period: Overall Study
Arm/Group | DTC Cohort | MTC Cohort
Started | 58 | 59
Completed | 58 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all participants who received at least one dose of the study drug and was the primary analysis set for efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | DTC Cohort | MTC Cohort | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (9.49) | 51.6 (14.11) | 56.2 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was the percentage of participants with best overall response (BOR) of complete response (CR) and partial response (PR) based on modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 for target lesions using magnetic resonance imaging/computed tomography (MRI/CT) scans, as determined by independent imaging review (IIR). CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter. ORR=CR+PR, was presented with 2-sided 95% confidence interval (CI) by the method of Clopper and Pearson.
Time Frame: From date of treatment start until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice to stop study treatment, or up to data cutoff date 11 April 2011, for up to approximately 2 years 5 months
Population: The Intent to Treat (ITT) Population included all participants who received at least one dose of the study drug and was the primary analysis set used for efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 58 | 59
Percentage of participants | 50.0 [36.6 to 63.4] | 35.6 [23.6 to 49.1]

2. Primary Outcome: Plasma Pharmacokinetics (PK): Steady State Area Under the Plasma Concentration Curve (AUC)
Description: Up to 9 samples per participant were obtained at specific time points. Plasma concentrations of lenvatinib were analyzed using standard analysis methods. Due to the sparse PK sampling in this study, the data were pooled with data from other Phase 1 studies conducted in participants with solid tumors for PK model development and covariate analysis. Individual exposure (steady state AUC) to lenvatinib in MTC and DTC subjects in this study was derived based on the individual predicted steady state AUC from the final PK model. Only data for participants taking 24 mg lenvatinib daily were reported (participants taking 20 mg lenvatinib daily were not included in this data set).
Time Frame: Cycle 1 Day 1 (predose and at 0.5 and 2 hours postdose), Cycle 1 Day 8 (predose), Cycle 2 Day 1 (predose and at 0.5 and 2 hours postdose), and Cycle 3 Day 1 (predose and at 2 hours postdose) (Cycle length= 28 days)
Population: PK population included all participants who received the 24 mg daily lenvatinib dose and had concentration values above the limit of quantification and non-missing PK sampling/dose time.
Measure: Median (Full Range); unit: ng·h/mL
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 47 | 56
ng·h/mL | 3840 [1610 to 6960] | 3350 [1040 to 6840]

3. Secondary Outcome: Change From Baseline in Free Thyroxine (T4)
Description: Blood samples to measure free T4 were collected at Screening (Baseline), Cycle 1 Day 15 (MTC cohort), Day 1 of Cycles 2 to 20, and Final Visit. Changes in free T4 concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included.
Time Frame: Day 1 or within 72 hours prior to Day 1 of Cycles 2 to 20, and Final Visit, up to data cutoff date 11 April 2011 (Cycle length= 28 days)
Population: All participants who received at least 1 dose of study drug. Only participants with both baseline and relevant visit/time point values were included. Data not reported for DTC cohort at Cycle 1 Day 15 and Cycle 20 Day 1 because no participant was evaluable at these time points.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 58 | 59
pmol/L
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 15 |  | -3.80
  Cycle 2 Day 1: number analyzed (Participants) | 53 | 57
  Cycle 2 Day 1 | -0.46 (5.149) | -0.86 (3.913)
  Cycle 3 Day 1: number analyzed (Participants) | 50 | 54
  Cycle 3 Day 1 | -0.92 (4.985) | -1.00 (4.028)
  Cycle 4 Day 1: number analyzed (Participants) | 48 | 50
  Cycle 4 Day 1 | -1.05 (5.581) | 0.34 (4.192)
  Cycle 5 Day 1: number analyzed (Participants) | 46 | 47
  Cycle 5 Day 1 | -1.03 (5.563) | -0.46 (3.878)
  Cycle 6 Day 1: number analyzed (Participants) | 43 | 45
  Cycle 6 Day 1 | -2.19 (5.373) | -0.17 (4.719)
  Cycle 7 Day 1: number analyzed (Participants) | 39 | 40
  Cycle 7 Day 1 | -2.32 (5.098) | -1.07 (5.403)
  Cycle 8 Day 1: number analyzed (Participants) | 37 | 37
  Cycle 8 Day 1 | -1.74 (5.504) | -1.13 (5.691)
  Cycle 9 Day 1: number analyzed (Participants) | 30 | 37
  Cycle 9 Day 1 | -0.39 (5.295) | 0.52 (5.213)
  Cycle 10 Day 1: number analyzed (Participants) | 30 | 32
  Cycle 10 Day 1 | -0.26 (6.397) | 1.33 (6.319)
  Cycle 11 Day 1: number analyzed (Participants) | 30 | 26
  Cycle 11 Day 1 | -0.27 (6.384) | 0.30 (5.551)
  Cycle 12 Day 1: number analyzed (Participants) | 30 | 21
  Cycle 12 Day 1 | -1.60 (6.331) | -0.43 (5.380)
  Cycle 13 Day 1: number analyzed (Participants) | 29 | 19
  Cycle 13 Day 1 | -0.09 (5.416) | 0.07 (4.347)
  Cycle 14 Day 1: number analyzed (Participants) | 27 | 14
  Cycle 14 Day 1 | -0.54 (5.772) | -0.82 (6.394)
  Cycle 15 Day 1: number analyzed (Participants) | 26 | 10
  Cycle 15 Day 1 | 0.63 (6.703) | -1.01 (5.505)
  Cycle 16 Day 1: number analyzed (Participants) | 24 | 9
  Cycle 16 Day 1 | -0.98 (7.150) | 0.60 (4.142)
  Cycle 17 Day 1: number analyzed (Participants) | 17 | 6
  Cycle 17 Day 1 | 1.20 (7.075) | 0.45 (3.528)
  Cycle 18 Day 1: number analyzed (Participants) | 10 | 6
  Cycle 18 Day 1 | 0.38 (4.648) | 2.17 (4.831)
  Cycle 19 Day 1: number analyzed (Participants) | 4 | 2
  Cycle 19 Day 1 | -0.65 (4.042) | 3.25 (4.596)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 20 Day 1 |  | 5.20
  Final Visit/Study Termination: number analyzed (Participants) | 21 | 22
  Final Visit/Study Termination | -0.36 (6.175) | 1.27 (4.584)

4. Secondary Outcome: Change From Baseline in Free Thyroid Stimulating Hormone (TSH)
Description: Blood samples to measure free TSH were collected at Screening (Baseline), Cycle 1 Day 15 (MTC cohort), Day 1 of Cycles 2 to 20, and Final Visit. Changes in free TSH concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included. For any free TSH result that was reported as <0.008 mIU/L, 0.004 mIU/L was used for calculating summary statistics.
Time Frame: as for outcome 3
Population: All participants who received at least 1 dose of study drug. For each change from baseline assessment time point, only participants with both baseline and relevant visit/time point values were included. Data not reported for DTC cohort at Cycle 1 Day 15 and Cycle 20 Day 1 because no participant was evaluable at these time points.
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 58 | 59
mIU/L
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 15 |  | 2.8030
  Cycle 2 Day 1: number analyzed (Participants) | 41 | 55
  Cycle 2 Day 1 | 0.4779 (3.07666) | 4.1585 (7.34946)
  Cycle 3 Day 1: number analyzed (Participants) | 38 | 52
  Cycle 3 Day 1 | 0.5161 (2.79122) | 5.5788 (13.76600)
  Cycle 4 Day 1: number analyzed (Participants) | 37 | 48
  Cycle 4 Day 1 | 0.6296 (2.29420) | 2.8751 (6.50098)
  Cycle 5 Day 1: number analyzed (Participants) | 35 | 45
  Cycle 5 Day 1 | 0.5024 (2.22721) | 3.7098 (6.60386)
  Cycle 6 Day 1: number analyzed (Participants) | 32 | 44
  Cycle 6 Day 1 | 0.8603 (3.09079) | 3.9822 (10.65477)
  Cycle 7 Day 1: number analyzed (Participants) | 30 | 40
  Cycle 7 Day 1 | 0.6660 (2.08608) | 8.4308 (22.51715)
  Cycle 8 Day 1: number analyzed (Participants) | 30 | 37
  Cycle 8 Day 1 | 0.2118 (3.16324) | 11.4131 (32.65896)
  Cycle 9 Day 1: number analyzed (Participants) | 25 | 37
  Cycle 9 Day 1 | 0.1270 (3.53020) | 6.6620 (18.89412)
  Cycle 10 Day 1: number analyzed (Participants) | 26 | 32
  Cycle 10 Day 1 | -0.3277 (2.87114) | 6.1934 (17.99762)
  Cycle 11 Day 1: number analyzed (Participants) | 25 | 26
  Cycle 11 Day 1 | -0.2940 (3.28192) | 2.7928 (9.42343)
  Cycle 12 Day 1: number analyzed (Participants) | 25 | 21
  Cycle 12 Day 1 | 0.3500 (5.43946) | 5.1879 (14.81415)
  Cycle 13 Day 1: number analyzed (Participants) | 25 | 19
  Cycle 13 Day 1 | -0.2799 (3.31518) | 2.0983 (7.03903)
  Cycle 14 Day 1: number analyzed (Participants) | 23 | 14
  Cycle 14 Day 1 | -0.6232 (3.09954) | 9.6490 (32.48910)
  Cycle 15 Day 1: number analyzed (Participants) | 22 | 10
  Cycle 15 Day 1 | -0.5911 (3.21447) | 0.9955 (4.93549)
  Cycle 16 Day 1: number analyzed (Participants) | 20 | 9
  Cycle 16 Day 1 | -0.3396 (3.68903) | 0.2971 (3.33103)
  Cycle 17 Day 1: number analyzed (Participants) | 14 | 7
  Cycle 17 Day 1 | -1.0352 (3.92286) | 7.4624 (16.18545)
  Cycle 18 Day 1: number analyzed (Participants) | 8 | 6
  Cycle 18 Day 1 | 0.0331 (0.24520) | 4.1232 (7.01461)
  Cycle 19 Day 1: number analyzed (Participants) | 4 | 2
  Cycle 19 Day 1 | 0.7805 (1.87674) | -0.2080 (0.29698)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 20 Day 1 |  | 0.0000
  Final Visit/Study Termination: number analyzed (Participants) | 17 | 20
  Final Visit/Study Termination | 1.0281 (2.07161) | 3.4905 (7.39625)

5. Secondary Outcome: Percent Change From Baseline in Concentrations of Thyroglobulin (DTC Only)
Description: Blood samples to obtain serum were collected at Cycle 1 Day 1 (Baseline), Day 1 of Cycles 2 to 19, Final Visit, and were analyzed for thyroglobulin concentration. Percent changes in thyroglobulin concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included.
Time Frame: Day 1 or within 72 hours prior to Day 1 of Cycles 2 to 19, and Final Visit, up to data cutoff date 11 April 2011 (Cycle length= 28 days)
Population: All participants who received at least 1 dose of study drug. For each change from baseline assessment time point, only participants with both baseline and relevant visit/time point values were included.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DTC Cohort
Number analyzed (Participants) | 52
percent change
  Cycle 2 Day 1: number analyzed (Participants) | 47
  Cycle 2 Day 1 | -62.21 (39.997)
  Cycle 3 Day 1: number analyzed (Participants) | 44
  Cycle 3 Day 1 | -77.80 (22.278)
  Cycle 4 Day 1: number analyzed (Participants) | 41
  Cycle 4 Day 1 | -79.25 (26.639)
  Cycle 5 Day 1: number analyzed (Participants) | 40
  Cycle 5 Day 1 | -76.00 (25.085)
  Cycle 6 Day 1: number analyzed (Participants) | 40
  Cycle 6 Day 1 | -20.36 (373.190)
  Cycle 7 Day 1: number analyzed (Participants) | 30
  Cycle 7 Day 1 | -73.38 (45.489)
  Cycle 8 Day 1: number analyzed (Participants) | 29
  Cycle 8 Day 1 | -79.96 (27.461)
  Cycle 9 Day 1: number analyzed (Participants) | 21
  Cycle 9 Day 1 | -73.98 (31.366)
  Cycle 10 Day 1: number analyzed (Participants) | 26
  Cycle 10 Day 1 | -78.26 (25.524)
  Cycle 11 Day 1: number analyzed (Participants) | 28
  Cycle 11 Day 1 | -75.54 (37.327)
  Cycle 12 Day 1: number analyzed (Participants) | 26
  Cycle 12 Day 1 | -73.51 (46.397)
  Cycle 13 Day 1: number analyzed (Participants) | 26
  Cycle 13 Day 1 | -74.05 (37.091)
  Cycle 14 Day 1: number analyzed (Participants) | 24
  Cycle 14 Day 1 | -78.70 (17.348)
  Cycle 15 Day 1: number analyzed (Participants) | 23
  Cycle 15 Day 1 | -80.28 (16.029)
  Cycle 16 Day 1: number analyzed (Participants) | 22
  Cycle 16 Day 1 | -76.38 (27.736)
  Cycle 17 Day 1: number analyzed (Participants) | 15
  Cycle 17 Day 1 | -62.99 (38.740)
  Cycle 18 Day 1: number analyzed (Participants) | 9
  Cycle 18 Day 1 | -72.67 (27.226)
  Cycle 19 Day 1: number analyzed (Participants) | 4
  Cycle 19 Day 1 | -50.65 (46.900)
  Final Visit/Study Termination: number analyzed (Participants) | 1
  Final Visit/Study Termination | -68.60

6. Secondary Outcome: Percent Change From Baseline in Concentrations of Calcitonin (MTC Only)
Description: Blood samples to obtain serum were collected at Cycle 1 Day 1(Baseline), Day 1 of Cycles 2 to 20, Final Visit, and were analyzed for calcitonin concentration. Percent changes in calcitonin concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MTC Cohort
Number analyzed (Participants) | 53
percent change
  Cycle 2 Day 1: number analyzed (Participants) | 51
  Cycle 2 Day 1 | -42.27 (38.754)
  Cycle 3 Day 1: number analyzed (Participants) | 47
  Cycle 3 Day 1 | -48.11 (30.976)
  Cycle 4 Day 1: number analyzed (Participants) | 44
  Cycle 4 Day 1 | -44.54 (38.794)
  Cycle 5 Day 1: number analyzed (Participants) | 40
  Cycle 5 Day 1 | -49.97 (34.634)
  Cycle 6 Day 1: number analyzed (Participants) | 39
  Cycle 6 Day 1 | -41.73 (46.653)
  Cycle 7 Day 1: number analyzed (Participants) | 34
  Cycle 7 Day 1 | -38.18 (62.721)
  Cycle 8 Day 1: number analyzed (Participants) | 33
  Cycle 8 Day 1 | -47.29 (46.101)
  Cycle 9 Day 1: number analyzed (Participants) | 29
  Cycle 9 Day 1 | -37.52 (72.588)
  Cycle 10 Day 1: number analyzed (Participants) | 29
  Cycle 10 Day 1 | -39.57 (60.118)
  Cycle 11 Day 1: number analyzed (Participants) | 24
  Cycle 11 Day 1 | -42.68 (61.797)
  Cycle 12 Day 1: number analyzed (Participants) | 19
  Cycle 12 Day 1 | -29.25 (105.440)
  Cycle 13 Day 1: number analyzed (Participants) | 17
  Cycle 13 Day 1 | -36.26 (89.612)
  Cycle 14 Day 1: number analyzed (Participants) | 12
  Cycle 14 Day 1 | -18.16 (148.928)
  Cycle 15 Day 1: number analyzed (Participants) | 9
  Cycle 15 Day 1 | -65.26 (24.553)
  Cycle 16 Day 1: number analyzed (Participants) | 8
  Cycle 16 Day 1 | -64.24 (30.394)
  Cycle 17 Day 1: number analyzed (Participants) | 7
  Cycle 17 Day 1 | -66.03 (23.777)
  Cycle 18 Day 1: number analyzed (Participants) | 6
  Cycle 18 Day 1 | -64.57 (27.982)
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | -44.30 (18.668)
  Cycle 20 Day 1: number analyzed (Participants) | 1
  Cycle 20 Day 1 | -29.40
  Final Visit/Study Termination: number analyzed (Participants) | 4
  Final Visit/Study Termination | -36.70 (28.296)

7. Secondary Outcome: Percent Change From Baseline in Concentrations of Carcinoembryonic Antigen (CEA) (MTC Only)
Description: Blood samples were collected at Cycle 1 Day 1(Baseline), Day 1 of Cycles 2 to 20, Final Visit, and were analyzed for CEA concentration. Percent changes in CEA concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MTC Cohort
Number analyzed (Participants) | 55
percent change
  Cycle 2 Day 1: number analyzed (Participants) | 54
  Cycle 2 Day 1 | -26.07 (45.864)
  Cycle 3 Day 1: number analyzed (Participants) | 49
  Cycle 3 Day 1 | -37.68 (42.236)
  Cycle 4 Day 1: number analyzed (Participants) | 46
  Cycle 4 Day 1 | -41.49 (48.035)
  Cycle 5 Day 1: number analyzed (Participants) | 42
  Cycle 5 Day 1 | -44.62 (42.138)
  Cycle 6 Day 1: number analyzed (Participants) | 42
  Cycle 6 Day 1 | -41.91 (47.388)
  Cycle 7 Day 1: number analyzed (Participants) | 36
  Cycle 7 Day 1 | -41.39 (45.677)
  Cycle 8 Day 1: number analyzed (Participants) | 34
  Cycle 8 Day 1 | -42.89 (47.818)
  Cycle 9 Day 1: number analyzed (Participants) | 30
  Cycle 9 Day 1 | -49.31 (32.185)
  Cycle 10 Day 1: number analyzed (Participants) | 30
  Cycle 10 Day 1 | -47.35 (31.621)
  Cycle 11 Day 1: number analyzed (Participants) | 25
  Cycle 11 Day 1 | -51.75 (29.671)
  Cycle 12 Day 1: number analyzed (Participants) | 20
  Cycle 12 Day 1 | -49.91 (32.597)
  Cycle 13 Day 1: number analyzed (Participants) | 18
  Cycle 13 Day 1 | -46.44 (35.967)
  Cycle 14 Day 1: number analyzed (Participants) | 13
  Cycle 14 Day 1 | -47.98 (38.324)
  Cycle 15 Day 1: number analyzed (Participants) | 10
  Cycle 15 Day 1 | -56.62 (34.051)
  Cycle 16 Day 1: number analyzed (Participants) | 9
  Cycle 16 Day 1 | -59.83 (34.762)
  Cycle 17 Day 1: number analyzed (Participants) | 7
  Cycle 17 Day 1 | -53.80 (37.981)
  Cycle 18 Day 1: number analyzed (Participants) | 6
  Cycle 18 Day 1 | -46.00 (39.905)
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | -45.65 (18.738)
  Cycle 20 Day 1: number analyzed (Participants) | 1
  Cycle 20 Day 1 | -61.40
  Final Visit/Study Termination: number analyzed (Participants) | 4
  Final Visit/Study Termination | -29.43 (31.453)

8. Secondary Outcome: Change From Baseline in Concentrations of Cytochrome C (CytoC)
Description: Blood samples to obtain serum were collected at Cycle 1 Day 1(Baseline), Cycle 1 Day 8, Cycle 2 Days 1,8 &15, Cycles 3 to 9,11,13 Day 1, Final Visit, and analyzed for CytoC concentration. Changes in CytoC concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included. For results reported as below quantifiable level (BQL), zero was used for calculating summary statistics. If more than 50% of the results at a visit were BQL, then only 'n', 'minimum' and 'maximum' were calculated for summary statistics.
Time Frame: Cycle 1 (Day 8), Cycle 2 (Days 1, 8 and 15), Cycles 3, 4, 5, 6, 7, 8, 9, 11, & 13 (Day 1), and Final Visit, up to data cutoff date 11 April 2011 (Cycle length= 28 days)
Population: All participants who received at least 1 dose of study drug. Only participants with both baseline and relevant visit/time point values were included. Data not reported for DTC cohort at Cycle 2 Day 1, for MTC cohort at Cycle 2 Day 15, Day 1 of Cycle 11 and 13 because no participant was evaluable at these time points.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 52 | 54
pg/mL
  Cycle 1 Day 8: number analyzed (Participants) | 52 | 52
  Cycle 1 Day 8 | 155.57 (825.091) | 502.84 (2146.291)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 2 Day 1 |  | 1679.40
  Cycle 2 Day 8: number analyzed (Participants) | 46 | 49
  Cycle 2 Day 8 | -218.45 (591.217) | 374.46 (2279.207)
  Cycle 2 Day 15: number analyzed (Participants) | 1 | 0
  Cycle 2 Day 15 | -215.50 |
  Cycle 3 Day 1: number analyzed (Participants) | 44 | 47
  Cycle 3 Day 1 | -175.43 (435.635) | 311.85 (2363.970)
  Cycle 4 Day 1: number analyzed (Participants) | 19 | 17
  Cycle 4 Day 1 | 1.38 (268.354) | 63.01 (1738.149)
  Cycle 5 Day 1: number analyzed (Participants) | 15 | 13
  Cycle 5 Day 1 | -21.32 (85.469) | 1078.85 (3793.235)
  Cycle 6 Day 1: number analyzed (Participants) | 14 | 10
  Cycle 6 Day 1 | 721.58 (1234.215) | 1411.29 (3855.502)
  Cycle 7 Day 1: number analyzed (Participants) | 10 | 7
  Cycle 7 Day 1 | 858.05 (1383.962) | 2184.30 (4689.181)
  Cycle 8 Day 1: number analyzed (Participants) | 10 | 5
  Cycle 8 Day 1 | 1358.51 (1364.706) | 451.36 (254.305)
  Cycle 9 Day 1: number analyzed (Participants) | 6 | 5
  Cycle 9 Day 1 | 1356.40 (913.685) | 459.38 (1572.717)
  Cycle 11 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 11 Day 1 | 139.60 |
  Cycle 13 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 13 Day 1 | 129.60 |
  Final Visit/Study Termination: number analyzed (Participants) | 19 | 23
  Final Visit/Study Termination | 249.31 (765.148) | -45.97 (1294.476)

9. Secondary Outcome: Change From Baseline in Concentrations of M-30 Neo-Antigen
Description: Blood samples to obtain serum were collected at Cycle 1 Day 1(Baseline), Cycle 1 Day 8, Cycle 2 Days 1,8 &15, Cycles 3 to 9,11,13 Day 1, Final Visit, and analyzed for M-30 concentration. Changes in M-30 concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included. For results reported as BQL, zero was used for calculating summary statistics. If more than 50% of the results at a visit were BQL, then only 'n', 'minimum' and 'maximum' were calculated for summary statistics.
Time Frame: Cycle 1 (Day 8), Cycle 2 (Days 1, 8 & 15), Cycles 3, 4, 5, 6, 7, 8, 9, 11 & 13 (Day 1) and Final Visit, up to data cutoff date 11 April 2011 (Cycle length= 28 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 52 | 54
U/L
  Cycle 1 Day 8: number analyzed (Participants) | 52 | 52
  Cycle 1 Day 8 | -5.22 (108.639) | 46.32 (197.509)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 2 Day 1 |  | -77.80
  Cycle 2 Day 8: number analyzed (Participants) | 46 | 49
  Cycle 2 Day 8 | -26.41 (257.723) | -49.33 (289.525)
  Cycle 2 Day 15: number analyzed (Participants) | 1 | 0
  Cycle 2 Day 15 | 35.30 |
  Cycle 3 Day 1: number analyzed (Participants) | 44 | 47
  Cycle 3 Day 1 | 19.70 (296.010) | -90.21 (314.343)
  Cycle 4 Day 1: number analyzed (Participants) | 19 | 17
  Cycle 4 Day 1 | -7.89 (336.124) | -97.53 (296.832)
  Cycle 5 Day 1: number analyzed (Participants) | 15 | 13
  Cycle 5 Day 1 | -24.83 (397.337) | -161.36 (265.548)
  Cycle 6 Day 1: number analyzed (Participants) | 14 | 10
  Cycle 6 Day 1 | -99.30 (321.554) | -161.30 (214.299)
  Cycle 7 Day 1: number analyzed (Participants) | 10 | 7
  Cycle 7 Day 1 | -168.50 (378.071) | -52.79 (129.671)
  Cycle 8 Day 1: number analyzed (Participants) | 10 | 5
  Cycle 8 Day 1 | -180.22 (386.682) | -92.44 (57.828)
  Cycle 9 Day 1: number analyzed (Participants) | 6 | 5
  Cycle 9 Day 1 | -111.92 (189.411) | -85.22 (161.751)
  Cycle 11 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 11 Day 1 | 55.00 |
  Cycle 13 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 13 Day 1 | -263.50 |
  Final Visit/Study Termination: number analyzed (Participants) | 19 | 23
  Final Visit/Study Termination | -151.73 (322.159) | -158.99 (355.903)

10. Secondary Outcome: Change From Baseline in Concentrations of Activated Caspase 3/7 (Casp 3/7)
Description: Blood samples to obtain serum were collected at Cycle 1 Day 1 (Baseline), Cycle 1 Day 8, Cycle 2 Days 1, 8, and 15, Cycles 3 to 9, 11, 13 (Day 1), Final Visit, and analyzed for Casp 3/7 concentration. Changes in Casp 3/7 concentration values from baseline to specific time points were calculated. Only participants with both baseline and relevant visit values were included. The concentrations of Casp 3/7 were BQL for most participants at most time points. For results reported as BQL, zero was used for calculating summary statistics. If more than 50% of the results at a visit were BQL, then only 'n', 'minimum' and 'maximum' were calculated for summary statistics.
Time Frame: Cycle 1 (Day 8), Cycle 2 (Days 1, 8, & 15), Cycles 3, 4, 5, 6, 7, 8, 9, 11, & 13 (Day 1) and Final Visit, up to data cutoff date 11 April 2011 (Cycle length= 28 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/W
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 58 | 59
U/W
  Cycle 1 Day 8: number analyzed (Participants) | 50 | 52
  Cycle 1 Day 8 | NA (NA) — BQL therefore not calculated | 0.0030 (0.00610)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 2 Day 1 |  | 0.0080
  Cycle 2 Day 8: number analyzed (Participants) | 44 | 49
  Cycle 2 Day 8 | NA (NA) — BQL therefore not calculated | 0.0039 (0.00822)
  Cycle 2 Day 15: number analyzed (Participants) | 1 | 0
  Cycle 2 Day 15 | 0.0110 |
  Cycle 3 Day 1: number analyzed (Participants) | 42 | 47
  Cycle 3 Day 1 | NA (NA) — BQL therefore not calculated | 0.0026 (0.00691)
  Cycle 4 Day 1: number analyzed (Participants) | 18 | 17
  Cycle 4 Day 1 | NA (NA) — BQL therefore not calculated | 0.0019 (0.00743)
  Cycle 5 Day 1: number analyzed (Participants) | 15 | 13
  Cycle 5 Day 1 | NA (NA) — BQL therefore not calculated | 0.0042 (0.00666)
  Cycle 6 Day 1: number analyzed (Participants) | 14 | 10
  Cycle 6 Day 1 | 0.0046 (0.00605) | NA (NA) — BQL therefore not calculated
  Cycle 7 Day 1: number analyzed (Participants) | 10 | 7
  Cycle 7 Day 1 | 0.0058 (0.00496) | 0.0044 (0.00692)
  Cycle 8 Day 1: number analyzed (Participants) | 10 | 5
  Cycle 8 Day 1 | 0.0078 (0.00771) | NA (NA) — BQL therefore not calculated
  Cycle 9 Day 1: number analyzed (Participants) | 6 | 5
  Cycle 9 Day 1 | 0.0067 (0.00480) | 0.0068 (0.01329)
  Cycle 11 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 11 Day 1 | NA (NA) — BQL therefore not calculated |
  Cycle 13 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 13 Day 1 | NA (NA) — BQL therefore not calculated |
  Final Visit/Study Termination: number analyzed (Participants) | 18 | 23
  Final Visit/Study Termination | NA (NA) — BQL therefore not calculated | NA (NA) — BQL therefore not calculated

11. Secondary Outcome: Duration of Response (DoR) Assessed as Per Independent Imaging Reviewers (IIR)
Description: DoR was based on IIR was the time from date of the first CR or PR until the date of first documentation of disease progression or date of death, if death occurred prior to disease progression, for the participants who had BOR of CR or PR. Participants without progressive disease or death were censored at the date of last adequate tumor assessment. Duration of response = End Date - Date of first CR or PR + 1
Time Frame: From date of the first CR or PR until the date of first documentation of disease progression or date of death, assessed up to data cutoff date 11 April 2011
Population: ITT population. Participants who were evaluable for this given measure at a given time point were included for this assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 29 | 21
Months | 12.7 [8.8 to NA] — Upper limit of confidence interval could not be calculated because of high number of participants that were censored from the analysis. | NA [5.7 to NA] — Data could not be calculated since less than 50 percent (%) of population had the event.

12. Secondary Outcome: Disease Control Rate (DCR) Assessed as Per IIR
Description: DCR was the percentage of the participants who had BOR of CR, PR, and stable disease (SD) with the minimum duration of SD lasting greater than or equal to 7 weeks, based on assessments by IIR. DCR = CR+PR+SD greater than or equal to 7 weeks
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 54 | 47
Percentage of participants | 93.1 [83.3 to 98.1] | 79.7 [67.2 to 89.0]

13. Secondary Outcome: Clinical Benefit Rate (CBR) Assessed as Per IIR
Description: CBR was the percentage of the participants who had BOR of CR, PR, and SD with the minimum duration of SD lasting greater than or equal to 23 weeks, based on assessments by IIR. CBR = CR+PR+SD greater than or equal to 23 weeks
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 45 | 38
Percentage of participants | 77.6 [64.7 to 87.5] | 64.4 [50.9 to 76.4]

14. Secondary Outcome: Time to Response (TTR) Assessed as Per IIR
Description: TTR was defined as "time from start of treatment to the time when a participant first achieves a response of PR/CR" based on assessments by IIR. TTR was only calculated for participants with confirmed PR or CR.
Time Frame: From date of treatment start until date of first CR or PR, assessed up to data cutoff date 11 April 2011
Population: The Efficacy Evaluable Population included all participants who received at least one dose of the study treatment, had a baseline and at least one posttreatment tumor response evaluation. Participants who were evaluable for this given measure at a given time point were included for this assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 28 | 19
Months | 3.6 [1.8 to 3.7] | 3.5 [1.9 to 3.7]

15. Secondary Outcome: Progression Free Survival (PFS) Assessed as Per IIR
Description: PFS was defined as the time from the date of treatment start until progressive disease or death from any cause in the absence of progressive disease. Disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions (taking as reference the smallest sum on study), recorded since the treatment started or the appearance of 1 or more new lesions as assessed by IIR using RECIST 1.0. The duration of PFS was calculated as end date minus date of first drug plus 1, based on assessments by IIR. PFS was calculated using Kaplan-Meier estimate and presented with 2-sided 95% Cl.
Time Frame: From date of treatment start until date of progressive disease or death from any cause, assessed up to data cutoff date 11 April 2011, for up to approximately 2 years 5 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 58 | 59
Months | 12.6 [9.9 to 16.1] | 9.0 [7.0 to NA] — Upper limit of confidence interval could not be calculated because of high number of participants that were censored from the analysis.

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of treatment start until death from any cause. The duration of OS was calculated as 'end date minus date of first drug plus 1', based on assessments by IIR. Participants without a reported death or those lost to follow-up were censored at their last known alive date at the database cutoff. OS was calculated using Kaplan-Meier estimate and presented with 2-sided 95% Cl.
Time Frame: From date of treatment start until date of death from any cause, assessed up to data cutoff date 11 April 2011, for up to approximately 2 years 5 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 58 | 59
Months | 27.7 [27.7 to NA] — Upper limit of confidence interval could not be calculated because of high number of participants that were censored from the analysis. | 16.6 [16.4 to NA] — Upper limit of confidence interval could not be calculated because of high number of participants that were censored from the analysis.

17. Secondary Outcome: Number of Participants With Non-Serious Adverse Events (AEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Lenvatinib
Description: Safety assessments consisted of monitoring and recording all AEs (serious and non-serious) and SAEs; concomitant medications, regular monitoring of hematology, blood chemistry, and urine values; periodic measurement of vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, New York Heart Association (NYHA) assessments, electrocardiograms (ECGs), echocardiograms; and performance of physical examinations.
Time Frame: For each participant, from the first dose till 30 days after the last dose of study treatment (up to approximately 10 years 4 months)
Population: Safety population included all participants who received at least 1 dose of study drug and had at least 1 posttreatment safety assessment.
Measure: Number; unit: Participants
Arm/Group | DTC Cohort | MTC Cohort
Number analyzed (Participants) | 58 | 59
Participants
  Non-Serious AEs | 58 | 59
  SAEs | 32 | 42

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 30 days after the last dose of study treatment (up to approximately 10 years 4 months)
Arm/Group | DTC Cohort | MTC Cohort
All-Cause Mortality (participants affected / at risk) | 44/58 | 37/59
Serious Adverse Events (participants affected / at risk) | 32/58 | 42/59
Other Adverse Events (participants affected / at risk) | 58/58 | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTC Cohort (N=58) | MTC Cohort (N=59)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (7) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcitoninaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 4 (5)
Lung infection (Infections and infestations) | 0 (0) | 3 (4)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Hypertension (Vascular disorders) | 2 (4) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder enlargement (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Echocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreatic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oncologic complication (Infections and infestations) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (2)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTC Cohort (N=58) | MTC Cohort (N=59)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 5 (8)
Bradycardia (Cardiac disorders) | 5 (6) | 0 (0)
Tachycardia (Cardiac disorders) | 7 (7) | 7 (9)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 4 (4)
Lacrimation increased (Eye disorders) | 4 (4) | 1 (1)
Visual impairment (Eye disorders) | 3 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 8 (12) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 20 (31) | 19 (38)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 18 (33) | 18 (28)
Constipation (Gastrointestinal disorders) | 16 (23) | 17 (37)
Diarrhoea (Gastrointestinal disorders) | 40 (146) | 45 (242)
Dry mouth (Gastrointestinal disorders) | 21 (25) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 8 (10)
Dysphagia (Gastrointestinal disorders) | 14 (17) | 12 (16)
Faeces pale (Gastrointestinal disorders) | 3 (6) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (5) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (9) | 7 (11)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 4 (7)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 4 (7)
Glossitis (Gastrointestinal disorders) | 5 (5) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 9 (14) | 12 (17)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 5 (5) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 30 (70) | 30 (82)
Oesophagitis (Gastrointestinal disorders) | 4 (5) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 3 (3) | 8 (10)
Oral pain (Gastrointestinal disorders) | 7 (14) | 8 (11)
Stomatitis (Gastrointestinal disorders) | 19 (55) | 15 (22)
Toothache (Gastrointestinal disorders) | 5 (5) | 6 (7)
Vomiting (Gastrointestinal disorders) | 23 (83) | 25 (91)
Asthenia (General disorders) | 14 (36) | 6 (32)
Chills (General disorders) | 3 (4) | 3 (5)
Fatigue (General disorders) | 35 (97) | 33 (84)
Influenza like illness (General disorders) | 4 (4) | 6 (8)
Malaise (General disorders) | 0 (0) | 5 (6)
Mucosal inflammation (General disorders) | 6 (7) | 7 (8)
Oedema peripheral (General disorders) | 14 (20) | 8 (8)
Pain (General disorders) | 6 (6) | 3 (3)
Pyrexia (General disorders) | 15 (21) | 12 (17)
Temperature intolerance (General disorders) | 4 (4) | 4 (4)
Bronchitis (Infections and infestations) | 8 (8) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 4 (5) | 3 (5)
Influenza (Infections and infestations) | 6 (10) | 7 (9)
Laryngitis (Infections and infestations) | 1 (1) | 3 (4)
Localised infection (Infections and infestations) | 2 (2) | 4 (8)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 5 (10)
Oral candidiasis (Infections and infestations) | 0 (0) | 4 (5)
Pharyngitis (Infections and infestations) | 4 (5) | 4 (7)
Rhinitis (Infections and infestations) | 3 (4) | 3 (3)
Sinusitis (Infections and infestations) | 3 (5) | 6 (12)
Tooth abscess (Infections and infestations) | 4 (4) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 12 (13) | 12 (19)
Urinary tract infection (Infections and infestations) | 11 (15) | 8 (17)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (7)
Activated partial thromboplastin time prolonged (Investigations) | 6 (6) | 5 (5)
Alanine aminotransferase increased (Investigations) | 7 (17) | 9 (21)
Aspartate aminotransferase increased (Investigations) | 9 (15) | 9 (18)
Blood creatine phosphokinase increased (Investigations) | 4 (6) | 2 (3)
Blood creatinine increased (Investigations) | 3 (4) | 4 (11)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 1 (1)
Blood pressure increased (Investigations) | 3 (9) | 4 (4)
Blood thyroid stimulating hormone increased (Investigations) | 4 (4) | 13 (16)
Electrocardiogram QT prolonged (Investigations) | 4 (7) | 4 (5)
Weight decreased (Investigations) | 39 (125) | 29 (81)
Decreased appetite (Metabolism and nutrition disorders) | 32 (61) | 32 (74)
Dehydration (Metabolism and nutrition disorders) | 9 (10) | 6 (10)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 (15) | 2 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (13) | 6 (9)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 (22) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (21) | 12 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (8) | 7 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (51) | 21 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (34) | 14 (31)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (15)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (27) | 7 (11)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (6) | 4 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 14 (19)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 (33) | 17 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (29) | 14 (27)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (11) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (46) | 17 (43)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 10 (14) | 13 (15)
Dysgeusia (Nervous system disorders) | 12 (14) | 9 (13)
Headache (Nervous system disorders) | 27 (49) | 27 (59)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 11 (15)
Hypoaesthesia (Nervous system disorders) | 3 (5) | 4 (4)
Paraesthesia (Nervous system disorders) | 7 (8) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 5 (8)
Tremor (Nervous system disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (7) | 8 (9)
Depression (Psychiatric disorders) | 11 (11) | 5 (6)
Insomnia (Psychiatric disorders) | 13 (14) | 7 (9)
Dysuria (Renal and urinary disorders) | 3 (3) | 3 (3)
Haematuria (Renal and urinary disorders) | 5 (7) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 2 (3)
Proteinuria (Renal and urinary disorders) | 41 (195) | 38 (160)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (46) | 24 (38)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 25 (39) | 20 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (32) | 16 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (28) | 13 (21)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 8 (13)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (35) | 13 (25)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (14) | 11 (17)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (8)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (10)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (37) | 15 (45)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 10 (12) | 16 (28)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (7)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (5) | 6 (16)
Skin fissures (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 3 (6) | 3 (6)
Skin lesion (Skin and subcutaneous tissue disorders) | 7 (11) | 4 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7)
Hypertension (Vascular disorders) | 45 (108) | 31 (74)
Hypotension (Vascular disorders) | 14 (19) | 10 (19)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (9)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (4)
Ear pain (Ear and labyrinth disorders) | 3 (5) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (4)
Cataract (Eye disorders) | 3 (3) | 0 (0)
Vision blurred (Eye disorders) | 4 (4) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 3 (5) | 3 (3)
Tongue disorder (Gastrointestinal disorders) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 3 (3)
Local swelling (General disorders) | 0 (0) | 3 (4)
Peripheral swelling (General disorders) | 5 (11) | 4 (4)
Seasonal allergy (Immune system disorders) | 2 (2) | 4 (4)
Pneumonia (Infections and infestations) | 4 (6) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 3 (4)
Vaginal infection (Infections and infestations) | 3 (3) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (5) | 5 (12)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (4)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 3 (4)
Blood triglycerides increased (Investigations) | 1 (3) | 3 (5)
Blood urea increased (Investigations) | 5 (9) | 2 (2)
Blood urine present (Investigations) | 3 (4) | 0 (0)
Haemoglobin decreased (Investigations) | 5 (5) | 2 (3)
Platelet count decreased (Investigations) | 2 (7) | 3 (3)
Prothrombin time prolonged (Investigations) | 3 (3) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hyperglycaemia (Investigations) | 4 (13) | 6 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (8) | 3 (4)
Confusional state (Psychiatric disorders) | 1 (1) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (12)
Sinus headache (Nervous system disorders) | 3 (3) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other